CLINICAL TRIAL: NCT00455182
Title: Acupuncture for Pain Management After Hip or Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll subjects who were willing to be randomized to control group
Sponsor: HealthEast Care System (Other)
Collaborators: University of Minnesota (Other); Northwestern Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE 06 10 007
Record Dates: First submitted 2007-03-29; First posted 2007-04-03 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Pain; Postoperative Complications
Keywords: Acupuncture; Hip Arthroplasty; Knee Arthroplasty; Pain Management
MeSH Terms: conditions — Pain; Postoperative Complications; Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Standard medical care
  Interventions: Procedure: Standard medical care
- 2 (Experimental): Acupuncture
  Interventions: Procedure: Acupuncture
- 3 (Sham Comparator): Sham acupuncture
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Standard medical care plus a single true acupuncture treatment.The needles are strategically inserted into the scalp, trunk, arms or legs (not near the surgical site) and manipulated. The needles are withdrawn between 5 minutes and 30 minutes after insertion.
  Arms: 2
Procedure: Sham Acupuncture — Standard medical care plus sham acupuncture. A single treatment, using a maximum of 9 sham needles, which adhere to the skin but do not penetrate it. The sham needles are strategically placed on the scalp, trunk, arms or legs (not near the surgical site)
  Other Names: The Park Sham Device
  Arms: 3
Procedure: Standard medical care — Standard medical care at Woodwinds Hospital includes guided imagery, essential oils and massage.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether patients treated with acupuncture post-operatively following knee or hip arthroplasty achieve better pain control as measured by the Visual Analog Scale and pain medication use.

DETAILED DESCRIPTION:
The postoperative acute pain of hip or knee arthroplasty can decrease early postoperative rehabilitation if uncontrolled. This pain is commonly managed with medications, which can be associated with a variety of side effects, including sedation, confusion, and falls. These side effects are particularly common among the elderly, who undergo the majority of these procedures. Adding non-pharmacologic therapies for pain management that can decrease the use of medication during the early post-operative period following hip or knee arthroplasty would be beneficial to patient recovery.

According to the National Institutes of Health (NIH) Consensus Statement, acupuncture has shown promising results in some medical situations, such as the management of post-operative and chemotherapy induced nausea and vomiting, as well as in post-operative dental pain. While a recent study funded by the NIH National Center for Complementary and Alternative Medicine showed that acupuncture provides pain relief and improves function for people with osteoarthritis of the knee, studies involving acupuncture and arthroplasty are few.

Two recent studies in which acupuncture was used in patients who underwent arthroplasty showed mixed results. In a study of ear acupuncture for pain relief in hip arthroplasty, there was decreased use of pain medication in those receiving acupuncture; however, the pain intensity rating was the same in both the acupuncture and sham acupuncture control groups (Usichenko TI, Pain, 2005). In a study that involved a longer duration of acupuncture therapy following total knee arthroplasty, patients who were treated with acupuncture in addition to standard physiotherapy showed no difference in pain, stiffness, or function at the end of six weeks when compared to patients who received standard physiotherapy(van Arendonk N, Physiotherapy, 2004-Abstract only). Further studies are needed to assess the efficacy of acupuncture in the post-operative pain management of patients who have undergone hip or knee arthroplasty.

The purpose of this pilot study is to test the feasibility of conducting such a study in order to competitively apply for funding for a full clinical trial.

This study is a randomized, single-blind, controlled trial with acupuncture in the immediate post-operative period versus sham acupuncture or standard medical care at HealthEast Woodwinds Hospital in Woodbury, Minnesota. Ninety (90) patients scheduled for elective hip or knee arthroplasty will be recruited from Woodwinds Hospital and randomized to one of the three treatment groups in a 1:1:1 ratio (30 patients in each group). Patients in the acupuncture or sham acupuncture group will receive one treatment on postoperative day 1. Pain medication use will be recorded and pain intensity will be assessed using the Visual Analog Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Undergoing total hip or total knee arthroplasty
* Spinal anesthesia during surgery

Exclusion Criteria:

* Arthroplasty of contralateral limb within the past three months
* Medical condition, in judgement of examiner, that may preclude safe participation in protocol or prevents completion of the study
* General anesthesia
* Use of any investigational drug in the past 30 days
* Has received acupuncture in the past
* Currently participating in another interventional study
* Unwilling to be randomized
* Patients who request Healing Touch, another form of alternative treatment that is offered at Woodwinds Hospital.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity as measured by the Visual Analog Scale | Before and immediately following treatment
Pain medication use | before and after treatment

SECONDARY OUTCOMES:
Cost of pain treatment | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hoeffel, M.D., Principal Investigator — Summit Orthopedics
Locations (1):
- HealthEast Woodwinds Hospital, Woodbury, Minnesota, United States

REFERENCES:
- [Background] N van Arendonk. Does the inclusion of acupuncture improve pain and functional outcome following total knee arthroplasty? Physiotherapy 90:168, 2004.
- [Background] Gilbertson B, Wenner K, Russell LC. Acupuncture and arthroscopic acromioplasty. J Orthop Res. 2003 Jul;21(4):752-8. doi: 10.1016/S0736-0266(03)00028-7. PMID 12798078
- [Result] Usichenko TI, Dinse M, Hermsen M, Witstruck T, Pavlovic D, Lehmann C. Auricular acupuncture for pain relief after total hip arthroplasty - a randomized controlled study. Pain. 2005 Apr;114(3):320-327. doi: 10.1016/j.pain.2004.08.021. PMID 15777857